CLINICAL TRIAL: NCT00000536
Title: Sodium Sensitivity in African Americans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 79; R01HL046630 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Sodium, Dietary

INTERVENTIONS:
Behavioral: sodium, dietary

SUMMARY:
To compare the effects of two levels of dietary sodium on blood pressure in Black men and women, and to determine what factors predict the degree of response.

DETAILED DESCRIPTION:
BACKGROUND:

The study permitted a more precise estimate of the effects of sodium chloride on blood pressure in Blacks and a systematic examination of sodium sensitivity defined by various methods. The results had significance in answering questions about risk factors for blood pressure in Blacks and for defining sodium sensitivity.

DESIGN NARRATIVE:

Double-blind, two-period cross-over. All participants were given six weeks of intensive nutritional counseling to lower 24-hour urine sodium output from an estimated 165 mEq/24 hours at baseline to less than 140 mEq/24 hours. Only those participants who excreted less than 140 mEq /24 hours after six weeks of intensive dietary sodium intervention and had greater than 70 percent adherence to study capsules were eligible for randomization. Eligible subjects were assigned to one of two treatment sequences: 100 mEq of sodium chloride capsules per day during period one followed by placebo capsules during period two; placebo capsules during period one followed by 100 mEq of sodium chloride capsules per day during period two. The major endpoint was change in diastolic and systolic blood pressure. A number of other measures were carried out, including blood chemistries, glucose tolerance (glucose and insulin), insulin resistance, urinary kallikrein, serum renin, and plasma norepinephrine. Other major aims of the trial included testing general new diagnostic criteria for sodium sensitivity, examining predictors of sodium sensitivity, and examining how changes in sodium intake influenced change in specific metabolic parameters. The trial design incorporated careful control of the dietary changes and strict standardization of blood pressure measurement with a random-zero device. The study was extended through June 1997 on FY 1995 funds.

ELIGIBILITY:
No eligibility criteria

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1992-07; Study Completion 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: Richard Grimm, Jr. — University of Minnesota

REFERENCES:
- [Background] Flack JM, Grimm RH Jr, Staffileno BA, Dnsc, Elmer P, Yunis C, Hedquist L, Dudley A. New salt-sensitivity metrics: variability-adjusted blood pressure change and the urinary sodium-to-creatinine ratio. Ethn Dis. 2002 Winter;12(1):10-9. PMID 11913598
- [Derived] Saviano A, Petruzziello C, Riccioni ME, Di Pumpo M, Petrucci M, Brigida M, Zanza C, Candelli M, Franceschi F, Ojetti V. Lower Gastrointestinal Bleeding in the Emergency Department: High- Volume vs. Low-Volume Peg Bowel Preparation for Colonoscopy: A Randomized Trial. Rev Recent Clin Trials. 2023;18(1):76-81. doi: 10.2174/1574887117666220908152754. PMID 36089784